CLINICAL TRIAL: NCT03786263
Title: The Canadian Childhood Nephrotic Syndrome (CHILDNEPH) Project
Brief Title: CHILDNEPH The Canadian Childhood Nephrotic Syndrome Study
Acronym: CHILDNEPH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB13-0059
Record Dates: First submitted 2018-06-06; First posted 2018-12-26 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Nephrotic Syndrome in Children; Nephrotic Syndrome, Minimal Change; Nephrotic Syndrome，Idiopathic
MeSH Terms: conditions — Nephrosis, Lipoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Treatments for NS: Observation of children (between the ages of 1 and 17) who are diagnosed with Nephrotic Syndrome at their initial presentation, first or second relapse.
  Observation of children who receive Glucocorticoids to treat Nephrotic Syndrome.
  Observation of children who receive other drugs (Second Line Agents) for Nephrotic Syndrome.

SUMMARY:
CHILDNEPH is a pan-Canadian project to observe clinical care for children with nephrotic syndrome. Previous studies have indicated that there is wide practice variation in how health care providers treat this remitting and relapsing disease of childhood. The disease mechanism is not yet understood, and long-term use of steroids can affect children's health. This study involves assessment of routine clinical care and establishing a long-term patient registry for children with nephrotic syndrome.

DETAILED DESCRIPTION:
CHILDNEPH is an ongoing prospective longitudinal study of children with incident and prevalent nephrotic syndrome. Children are recruited from 12 centres across Canada and followed for at least 30 months. The project starting in August of 2013 with the goal of following 400 patients. Data is collected at enrollment, beginning and end of each relapse, semi-annual visits and end of study. Detailed prescription data is collected regarding glucocorticoids and all second line agents. All relapses are recorded with time to urinary remission of proteinuria.

The investigators are moving towards registry based trials to determine optimal treatment protocols for nephrotic syndrome with an overall goal to minimize glucocorticoid exposure, a patient priority.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with Nephrotic Sydrome at initial presentation, first or second relapse

Exclusion Criteria:

* unable to participate in English or French
* Nephrotic Syndrome is secondary to other disease
* Younger than one year old or older than 17 years

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (ages 1 to 17 years) who are diagnosed with Nephrotic Syndrome (minimal change disease or idiopathic NS) who present at a participating pediatric nephrology clinic in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-08-03 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Association of steroid dose prescribed with relapse rates | 30 months up to 90 months
  Total steroid dose prescribed per unit time is determined by the total dose patients are prescribed during observation divided by total number of days on treatment. Dose will always be in mg/m2 prednisone equivalents. The relapse rate is the number of relapses/per person unit time.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Samuel, MD, MSc, Principal Investigator — University of Calgary
Locations (12):
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, University of Alberta, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Winnipeg Children's Hospital, University of Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario (CHEO) University of Ottawa, Ottawa, Ontario
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - CHU Ste. Justine, Montreal, Quebec
  - Montreal Children's Hospital - McGill University, Montreal, Quebec
  - Royal University Hospital, University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2015-02-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03786263/Prot_000.pdf